CLINICAL TRIAL: NCT00220870
Title: Shared Decision Making in the Therapy of Schizophrenia
Brief Title: Shared Decision Making for Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 217-43794-5/9; 217-43794-5/9
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2010-04-08 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia
Keywords: schizophrenia; shared decision making; compliance; maintenance therapy
MeSH Terms: conditions — Schizophrenia; Patient Compliance | interventions — Decision Support Techniques

INTERVENTIONS:
Behavioral: Decision aid

SUMMARY:
The impact of a decision aid for inpatients with schizophrenia on perceived involvement and compliance is studied in comparison with routine care.

DETAILED DESCRIPTION:
to follow

ELIGIBILITY:
Inclusion Criteria:

* schizophrenia (ICD10)
* age 18 - 65 years
* inpatients

Exclusion Criteria:

* mental retardation
* no informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-01; Study Completion 2005-08

PRIMARY OUTCOMES:
Patients' compliance

SECONDARY OUTCOMES:
perceived involvement in medical decisions
rehospitalizations
QoL

CONTACTS AND LOCATIONS:
Overall Officials: Werner Kissling, MD, Study Chair — TU München, Psychiatric Department
Locations (1):
- Psychiatric Department, TU München, München, Germany

REFERENCES:
- See also: Related Info — http://www.patient-als-partner.de